CLINICAL TRIAL: NCT07340359
Title: Effect of Yellow Light AG Mobile Phone Screen on Dry Eye and Asthenopia.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2025-1513
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Digital Eye Strain; Computer Vision Syndrome; Dry Eye; Asthenopia
MeSH Terms: conditions — Dry Eye Syndromes; Asthenopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- yellow light AG group (Experimental): use yellow light AG smartphone
  Interventions: Behavioral: reading 2h on smartphone
- control group (Placebo Comparator): use non-yellow light AG smartphone
  Interventions: Behavioral: reading 2h on smartphone

INTERVENTIONS:
Behavioral: reading 2h on smartphone — reading 2h on smartphone

SUMMARY:
This study aimed to evaluate the protective effects of yellow-light etching anti-glare (AG) screen on Digital Eye Strain (DES) induced by prolonged video display terminal (VDT) use under dim environment, Based on the proved positive effect of the circular polarization (CP) screen, providing insights for new eye-protection strategy in the highly digital modern era. In a randomized, double-blind controlled trial, 70 eligible volunteers (diopter ≤ -6.0D; anisometropia ≤ 2.0D) were divided into AG+CP or CP only groups. Participants performed a 2-hour e-book reading task using assigned AG+CP or CP only smartphones. Subjects' severity of DES pre- and post-reading were evaluated from two aspects: the degree of dry eye symptoms and asthenopia. Dry eye symptoms indicators (OSDI, TMH, NIBUT, FBUT, CFS, Schirmer I Test) and asthenopia indicators (CVSS17, Bulbar redness, HFC) were measured and compared.

DETAILED DESCRIPTION:
The inclusion criteria required subjects to have myopia diopter not exceeding -6.00D, hyperopia not exceeding +2.0D, astigmatism not exceeding -2.00D, anisometropia between both eyes not exceeding 2.00D. The key exclusion criteria were as follows: (1) strabismus and amblyopia; (2) used eye drops within 1 week; (3) had undergone eye surgery within 6 months; (4) worn contact lenses within the last 2 weeks; (5) had serious eye discomfort in the last 7 days; (6) breastfeeding or pregnant women and patients with severe systemic diseases, psychosis or dementia. Subjects did not know the characteristics of the smartphones they use. The subjects were asked not to use video terminals such as mobile phones within 30 minutes before the study began.

Subjects were divided into 2 groups using AG+CP or CP only smartphone provided. During the whole experiment, subjects were in a room with 2 lux-environment illuminance, screen brightness about 10nit to mimic the situation before sleep. Light source stability (working surface illuminance fluctuation) greater than 99% during the whole experiment, desktop range uniformity greater than 80%. Indoor air conditioning control temperature: 22-25 degrees Celsius, humidity: 50-70%RH. Mobile phones were placed on a fixed holder (the angle and height of the phone holder can be adjusted to ensure the suitability of participants). All subjects' eyes were 40cm away from the mobile phone screen and seated on a chair of fixed position and appropriate height. Subjects were asked to finish 2-hour reading on the specific smartphone. Reading materials are downloaded in advance to the smartphone and presented using specific reading software and settings. During the study period, subjects were not allowed to do any behavior unrelated to watching the screen for a long time (more than 1 minute). All experiments were conducted between 8:00 and 11:00 to minimize the impact of electronic screen use during the day. Ocular surface disease index (OSDI), tear meniscus height (TMH), noninvasive tear break-up time (NIBUT), Fluorescein tear break-up time (FBUT), corneal fluorescein staining (CFS) and Schirmer I test were measured to evaluate the degree of dry eye symptom. Computer vision syndrome scale 17 (CVSS17), bulbar redness and high-frequency component of accommodative microfluctuations (HFC), were identified as assessment of asthenopia. The intervention and assessments were delivered both at before and after smartphone reading by qualified clinical ophthalmologists in a hospital setting.

ELIGIBILITY:
Inclusion Criteria:

* 1.have basic reading comprehension skills and to be older than 18 years old. 2.diopter of both eyes not exceeding -6.0D and anisometropia not exceeding 2.0D.

Exclusion Criteria:

* 1.presbyopia or decreased regulation function, 2.ocular inflammation and disease, 3.worn contact lens within 1 month, 4.history of eye surgery within 6 months, 5.lactating or pregnant woman, 6.have severe systemic diseases.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12-24 (Actual); Primary Completion 2026-01-22 (Estimated); Study Completion 2026-01-22 (Estimated)

PRIMARY OUTCOMES:
Flourescence tear break-up time | 1 month
  Drop a drop of physiological saline onto a sodium fluorescein test strip. Gently touch the middle of the conjunctiva of both lower eyelids of the examinee with the test strip respectively, and instruct the examinee to blink their eyes gently and look straight ahead. The examiner observed the tear film of the examinee with cobalt blue light under a slit lamp. The time of tear film rupture was the time from the examinee opening their eyes to the appearance of the first black spot on the tear film. Three TBUT tests were detected and recorded for each eye respectively, and the average and maximum values were taken.
HFC (high frequency component of accommodative fluctuation) | 1 month
  The SCR mode of the ACOMOREF K-MODEL computerized optometer was adopted. The subjects were asked to keep a close eye on the image. The image distance was gradually moved from infinity to 1m, 60cm, and 30cm, and remained at each of the four distances for 20 seconds. The equipment would analyze and record the high-frequency fluctuations of the subjects' ciliary muscles, known as HFC. After the test of the first eye, Take a 20-second break to test the second eye.
non-invasive tear break-up time | 1 month
  The Oculus ocular surface comprehensive analyzer was adopted. The examinees sat upright in front of the instrument and were asked to blink their eyes lightly and then look at the red marked object. The instrument automatically conducted ocular surface image analysis to obtain and record the first NIBUT and average NIBUT of the examinees

SECONDARY OUTCOMES:
tear meniscus height | 1 month
  The Oculus ocular surface comprehensive analyzer was used. The person being examined sat upright in front of the instrument and was asked to blink their eyes slightly and then look at the red marked object. The instrument automatically analyzed the ocular surface images to obtain the lacrimal river height data
corneal fluorescein staining | 1 month
  After character searching, gaming and video tasks utilizing specific smartphones for totally 45 minutes, CFS was measured.
computer vision symptom scale 17 | 1 month
  A subjective scale reflecting the symptoms of visual fatigue, including the occurrence frequency and intensity of 17 ocular and extraocular symptoms
Schirmer I test | 1 month
  The subjects were tested under non-anesthetic conditions. A 5mm×35mm filter paper was placed in the conjunctival sac of the inner 1/3 of the lower eyelid, with the remaining part hanging over the skin surface. The subjects were asked to gently close their eyes. After 5 minutes, the length of the filter paper soaked by tears was measured and recorded

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine (SAHZU), Hangzhou, Zhejiang, China